CLINICAL TRIAL: NCT00672009
Title: A Phase II Study of Ixabepilone Prior to Surgery for High-risk Localized Prostate Cancer
Brief Title: A Study of Ixabepilone Before Surgery for High-Risk Localized Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor terminated funding for the study.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Mitchell Gross, MD, PhD, Director of Research, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13963
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Prostatic Diseases; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male; Adenocarcinoma; Prostatic Neoplasms; Neoplasms, Glandular and Epithelial; Carcinoma
Keywords: prostate cancer; radical prostatectomy; ixabepilone
MeSH Terms: conditions — Prostatic Diseases; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male; Adenocarcinoma; Prostatic Neoplasms; Neoplasms, Glandular and Epithelial; Carcinoma | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One (Experimental)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Ixabepilone 35 mg/m^2 intravenously over 3 hours every 21 days for 4 cycles.
  Other Names: BMS-247550

SUMMARY:
The purpose of this research study is to determine the safety and effectiveness of the investigational drug, Ixabepilone, in men with high risk prostate cancer who plan to receive surgery.

Prostate cancer is a common and important health issue facing men in the United States. Most patients with prostate cancer are identified when the disease is limited to the prostate gland itself (localized prostate cancer). A standard treatment for some patients with localized prostate cancer is removal of the prostate gland in an operation known as a "radical prostatectomy." A sub-set of patients with localized prostate cancer can be identified who are at high-risk of suffering a recurrence of prostate cancer after radical prostatectomy. For these patients, additional treatments are being investigated to combine with surgery in the hopes of increasing the chances for cure.

Several kinds of chemotherapy medicines have been used for advanced prostate cancer which returns after initial therapy. Epothilones are a newly developed class of chemotherapy drugs that appear promising for the treatment of many forms of cancer. Ixabepilone is drug in the epothilone class of chemotherapy medicines that has shown encouraging results for the treatment of advanced prostate cancer and other cancers in clinical trials.

This trial will include men with high-risk localized prostate cancer who will receive treatment with ixabepilone (4 cycles over 12 weeks) prior to radical prostatectomy. The goal of this trial will be to determine if analysis of genes and proteins in prostate cancer tissue taken before and after treatment can be used to predict ixabepilone response. In addition, this trial will evaluate the safety and feasibility of administering ixabepilone prior to radical prostatectomy for patients at high-risk of developing recurrent prostate cancer.

The study has three phases: Screening, Treatment and Follow-up

* Screening: Eligibility will be verified
* Treatment: Subjects will receive Ixabepilone, which will be administered every 21 days for 4 cycles prior to surgery
* Follow up: Subjects will be followed every 6 months for up to 5 years.

In addition, tissue will be collected at the time of surgery for genetic and protein studies. Blood will also be collected pre and post therapy for proteomic and/or genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed localized prostate cancer
* Predicted probability of recurrence >/= 30% as defined by the updated Kattan nomogram
* Pathologic material available for gene expression analysis including cancer present in 2 or more cores and availability of unstained slides or formalin-fixed paraffin embedded tissue blocks.
* No prior prostate cancer therapy (including hormonal, chemotherapy, radiation or surgery)
* Subjects must be considered as candidates for radical prostatectomy
* EGOG status
* Men of child-bearing potential are required to use an effective means of contraception
* Required Initial Laboratory Values:
* ANC >/= 1500/uL
* Platelet Count >/= 100000/uL
* Creatinine Bilirubin AST < 2.5 X ULN
* ALT < 2.5 X ULN
* Hemoglobin >/= 9.0 g/dL

Exclusion Criteria:

* A history of significant ventricular arrhythmias
* Neuropathy (> grade 1)
* Recent (within 6 months) myocardial infarction, congestive heart failure, transient ischemic attack or stroke
* Active angina, including active stable and unstable angina
* Acute deep venous thrombosis and/or pulmonary embolism in the past 6 months
* Any prior hormonal therapy including the use of PC Spes or estrogen containing nutriceuticals
* Other co-existing malignancies or malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma.
* Patients with malignancy diagnosed more than 5 years ago and are disease free for at least 5 years are not excluded.
* Recent (within 4 weeks) surgery or incomplete healing from surgery
* Known history of hypersensitivity reaction to a drug formulated in Cremophor EL
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of trial treatment
* Active infection requiring antibiotic therapy, or serious intercurrent illness.
* Any other major illness that in the investigators judgment will substantially increase the risk associated with the subject's participation in this study.
* Unwillingness or inability to comply with procedures required in this protocol.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine the biochemical response rate (defined as >/= 50% reduction in PSA from baseline to the post-therapy value) for non-castrate patients with localized prostate cancer and a >/= 30% risk of recurrence within 5 years. | 4 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell E Gross, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States